CLINICAL TRIAL: NCT00585520
Title: Sex Differences in Progesterone Effects on Responses to Stress and Drug Cues
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Rajita Sinha, Professor, Yale University
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 0609001804; P50DA016556 (NIH)
Record Dates: First submitted 2007-12-25; First posted 2008-01-03 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-02

CONDITIONS: Cocaine Dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PG (Active Comparator)
  Interventions: Drug: Progesterone
- PLA (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Progesterone — 200mg BID for 5 days
  Arms: PG
Drug: Placebo — Placebo
  Arms: PLA

SUMMARY:
Cocaine dependence is a chronic, relapsing disorder in which stress/negative mood and exposure to drug-related stimuli or "cues" are associated with high rates of relapse (McKay et al., 1995; O'Brien et al., 1998; R. Sinha, 2001; Shaham et al., 2003). In particular, sex differences in relapse precipitants have been noted, with women reporting greater stress related relapses while men report higher number of relapses associated with drug cue/temptation situations (Lex, 1991; McKay et al., 1996; R. Sinha, 2001; R. Sinha, Rounsaville BJ, 2002). Current SCOR studies have shown that stress and cocaine cues increase drug craving and stress related arousal, responses that differ in cocaine men and women (R. Sinha et al., 2003; H.C. Fox et al., 2005a). Furthermore, stress-induced cocaine craving and HPA responses are predictive of cocaine relapse, which is also moderated by gender (R. Sinha et al., 2006). However, no previous research has examined the basis of sex differences in stress and cue induced craving and arousal, both of which are known to increase relapse susceptibility. Greater knowledge of the sex-specific neurobiology of cocaine dependence will facilitate development of gender-specific cocaine relapse prevention efforts.

Growing evidence supports a role for gonadal hormones in explaining the sex differences observed in stress responses as well as in the behavioral responses to cocaine (Festa & Quinones-Jenab, 2004; K. Carroll, Fenton LR, Ball SA, Nich C, Frankforter TL, Shi J, Rounsaville BJ, 2004; Lynch, 2006; Kajanti & Phillips, 2006). Estrogen increases behavioral responses to cocaine, while presence of progesterone decreases subjective and behavioral effects of cocaine, more so in females than males (Jackson et al., 2006; Sofuogu et al., 1999; M. Sofuoglu et al., 2002; Evans & Foltin, 2006). Stress and cocaine each enhance brain stress circuits, namely the corticotrophin releasing factor (CRF)-hypothalamic-pituitary-adrenal (HPA) axis and central noradrenergic/sympatho-adrenomedullary (SAM) pathways and both activate the mesolimbic dopaminergic systems involved in the rewarding effects of cocaine (ADD REFS). Exposure to Stress, cocaine or cocaine cues will each increase cocaine craving and HPA axis responses. Importantly, progesterone which affects behavioral responses to cocaine, also plays a key role in stress regulation. However, it is not known whether progesterone alters stress-induced and drug cue-induced craving and related stress arousal, markers that predict cocaine relapse outcomes. Our preliminary data suggest that women exposed to stress and to drug cues in the laboratory during the luteal phase (high progesterone) show lower stress induced and drug cue-induced craving, anxiety and cortisol responses compared to those in the late follicular phase (high estrogen) (see preliminary Studies section CX). On the basis of this previous research, we propose a double-blind placebo controlled study of to examine progesterone's effects on stress and cue-related responses in cocaine dependent men and women. We hypothesize that high dose of progesterone (200 mg bid) vs. placebo will alter stress-induced cocaine craving, negative affect, physiological and HPA responses to stress, and these changes will be greater in women than men.

ELIGIBILITY:
Inclusion Criteria:

* Female and males, aged 18 to 50 years
* Able to read and write
* Meet current DSM-IV criteria for cocaine dependence; and report current cocaine use of at least once a week or more; confirmation of cocaine use via positive urine test at initial assessment and upon inpatient admission.
* For women, regular menses every 25-35 days
* In good health as verified by medical history, screening examination, and screening laboratory tests
* For women, not pregnant as determined by pregnancy screening, nor breast feeding, and using acceptable birth control methods other than hormonal contraceptives

Exclusion Criteria:

* History of major medical illnesses; including liver diseases, abnormal vaginal bleeding, suspected or known malignancy, thrombophlebitis, deep vein thrombosis, pulmonary embolus, clotting or bleeding disorders, heart disease, diabetes, history of stroke or other medical conditions that the physician investigator deems as contraindicated for the patient to be in the study
* Regular use of psychotropic medication (antidepressants, antipsychotics, or anxiolytics) and recent psychiatric diagnosis and treatment for Axis I disorders including major depression, bipolar affective disorder, schizophrenia or panic disorder; Meet current criteria for dependence on another psychoactive substance, excluding nicotine and caffeine; Any current use of opiates or past history of opiate abuse/dependence.
* For women, amenorrhea
* Known allergy to progesterone or peanuts (vehicle for micronized progesterone).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2007-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
HPA responses to stress | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Rajita Sinha, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine: Research Program on Stress, Addiction, and Psychopathology, New Haven, Connecticut, United States